CLINICAL TRIAL: NCT00407446
Title: Long-Term Use of Sildenafil in the Therapeutic Management of Heart Failure
Brief Title: PDE5-Inhibition With Sildenafil in Chronic Heart Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Milan (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 124-04
Record Dates: First submitted 2006-12-01; First posted 2006-12-05 (Estimated); Last update posted 2006-12-14 (Estimated); Status verified 2006-12

CONDITIONS: Heart Failure
Keywords: PDE5 inhibition; chronic heart failure; endothelial function; exercise ventilation
MeSH Terms: conditions — Heart Failure | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: sildenafil

SUMMARY:
To test the hypothesis that long-term PDE5-inhibition by overexpressing the nitric oxide pathway is beneficial in chronic heart failure patients.

Double-blind and placebo-controlled trial. Primary end-points: quality of life and exercise performance

DETAILED DESCRIPTION:
In chronic heart failure (CHF), endothelial function (EF) deterioration and muscle underperfusion elicit ergoreflex exercise oversignaling, hyperventilation and breathlessness. PDE5 inhibition, by improving EF, might be beneficial. We tested this hypothesis in a long-term therapeutic trial. CHF patients were randomly assigned to placebo (23 cases, group 1) or sildenafil (23 cases, group 2) in addition to their current antifailure therapy, for 6 months. In group 2 and not in group 1, assessments at 3 and 6 months showed the following changes: reduction of systolic pulmonary artery pressure (-25.2 and -29.0 %), ergoreflex effect on ventilation (-66.6 and -72.5%), ventilation to CO2 production slope (VE/VCO2, -14.0 and -16.0%) and breathlessness (-29.6 and -27.1%); increase of brachial artery flow-mediated dilatation (FMD, +57.6 and +67.0%), peak exercise O2 uptake (peak VO2, +25.0 and +26.3%) and ratio of VO2 to work rate changes (VO2WR, +20.7 and +22.0%). These changes were significant at p<0.01. In group 2 and not in group 1, a significant correlation was found, at 3 and 6 months, between changes in FMD and those in ergoreflex VE. Changes in ergoreflex correlated with those in peak VO2 and VE/VCO2 slope. No remarkable side effects were noted, but flushing in 3 patients.

In CHF, benefits of sildenafil are sustained and consist of improvement in EF, modulation in ergoreflex signaling, attenuation in exercise hyperventilation and breathlessness, increase in aerobic efficiency and exercise performance. Thus, sildenafil can affect peripheral mechanisms of breathlessness and may be viewed as an effective and safe adjunct to the therapeutic armamentarium of CHF.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility criteria were: consent to participate in the study after detailed information about procedures, possible clinical benefits and risks; ability to complete a maximal exercise test; forced expiratory volume in 1 sec/forced vital capacity ratio>70%; left ventricular ejection fraction  45%, determined by echocardiography.

Exclusion Criteria:

* Patients were not recruited if they had systolic blood pressure > 140 and <110 mmHg, diabetes mellitus, therapy with nitrate preparations, history of sildenafil intolerance, significant lung or valvular diseases, neuromuscular disorders, exercise-induced myocardial ischemia, atrial fibrillation (6), claudication, peripheral vascular disease.

Ages: 30 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-01; Study Completion 2005-02

PRIMARY OUTCOMES:
Exercise performance, ventilation efficiency, symptoms

SECONDARY OUTCOMES:
quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Marco Guazzi, MD, Principal Investigator — University of Milano
Locations (1):
- Marco Guazzi, MD, PhD University of Milano, Milan, Italy

REFERENCES:
- [Background] Katz SD, Parker JD, Glasser DB, Bank AJ, Sherman N, Wang H, Sweeney M. Efficacy and safety of sildenafil citrate in men with erectile dysfunction and chronic heart failure. Am J Cardiol. 2005 Jan 1;95(1):36-42. doi: 10.1016/j.amjcard.2004.08.060. PMID 15619391